CLINICAL TRIAL: NCT03603301
Title: Vision in Children Born to Opioid-dependent Methadone-maintained Mothers
Acronym: VINCH
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Waterloo (Other)
Responsible Party: Sponsor
Other Study IDs: GN16OP130p
Record Dates: First submitted 2017-03-22; First posted 2018-07-27 (Actual); Last update posted 2018-08-01 (Actual); Status verified 2018-07

CONDITIONS: Vision Disorders; Strabismus; Nystagmus; Binocular Vision Disorder
MeSH Terms: conditions — Vision Disorders; Strabismus; Nystagmus, Pathologic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators will re-investigate 150 children studied extensively in the past. 100 of these children were born to mothers prescribed methadone during their pregnancy because of opiate dependency, and 50 were comparison children who were not exposed to drugs. These children were investigated when they were newborn babies, and again when they were six months old, and a quarter of the drug-exposed babies had problems with their eyesight, whilst very few of the comparison children has eyesight problems. The investigators would like to see whether the eyesight problems are still present in the children now that they are older. Because they are older, more detailed testing can be undertaken which will help to understand how drug exposure in the womb may have affected their eyesight. The investigators will recruit new, comparison children to the study to match the number of comparison children with the number of drug-exposed children. The findings will be relevant and important when advising mothers on drug use - both prescribed and illicit - when they are pregnant.

DETAILED DESCRIPTION:
Multiple researchers across the world over many decades have noted eyesight problems in children born to mothers who use drugs during pregnancy. From our earlier work on this group of children, we have detailed knowledge of which drugs each mother used, making this group of children uniquely important for understanding the consequences of drug use during pregnancy. Although methadone use in the UK is dropping as heroin misuse falls, there is currently an international epidemic of babies being born to mothers using illicit or prescribed opioid drugs (e.g. methadone, heroin, opiate-based painkillers). These babies may be at risk of the same eyesight problems as this Scottish cohort. Knowing the longer-term consequences and disseminating the findings to relevant international clinical groups could help to alleviate the consequential damage, through better information for mothers and through better and prompter management of affected children.

The study is planned to run for 2 years. It is anticipated that a maximum of 65 drug-exposed children (out of the original 100) will attend, and will therefore aim to also investigate 65 comparison children, as many as possible of whom will belong to the original cohort of 50 comparison children.

Testing will take place in the Children's Clinical Research Facility (CRF), on the campus of the Queen Elizabeth University Hospital and Royal Hospital for Children, Glasgow. A CRF paediatric nurse will recruit, coordinate and administrate the study. They will manage the child's progress through the assessment session, measure height, weight and head circumference, document demographic, social and educational details from the child's carer, and will apply two questionnaires to the carers. Eyesight tests will be done by a specialist paediatric orthoptist, and will include acuity (the smallest letter correctly identified), stereoacuity (perception of depth) and looking for squints or nystagmus (shaking or wobbling of the eyes).

Highly specialised eye tests (eye movement recordings and visual evoked potentials) will also be undertaken.

If any abnormalities are noted from these tests, the child will be given eyedrops to dilate their pupils. All children will be seen by a paediatric ophthalmologist who will look at the back of their eyes, and check whether they need glasses, or whether their glasses are correct. A medical history will be taken. If any problems are noted during the visit (e.g. visual, medical, social), the child will be referred to relevant services after discussion with their carer.

The data will be added to the existing database for these children, and the test results correlated with the results found at birth and at six months, and with the any known drug exposure of each child.

ELIGIBILITY:
Inclusion Criteria:

* cases: born to opioid-dependent mothers prescribed substitute methadone during pregnancy and delivered after 36 completed weeks' gestation.
* comparisons: healthy, non drug-exposed infants delivered within the same maternity unit, matched for gestation, birthweight ± 250g and Carstairs deprivation score ± 1; attempted match for smoking

Exclusion Criteria:

* congenital ocular abnormality; significant neonatal illness

Ages: 7 Years to 10 Years | Sex: All
Age Groups: Child
Study Population: 100 drug-exposed neonates and 50 comparison infants, all born between 13/08/2008 and 30/04/2009 at the Princess Royal Maternity in Glasgow, previously recruited to the VIDI study; an additional 50 classroom comparison children.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-02 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
presence of strabismus, nystagmus, reduced acuity, significant refractive error | 2 years
  natural history of visual abnormalities following in utero exposure to methadone +/- other drugs

SECONDARY OUTCOMES:
correlation of abnormality or normality with prenatal drug exposure | 2 years
  to map visual findings to the known prenatal drug exposure and infant visual findings for each child

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Hamilton, PhD, Principal Investigator — NHS Greater Glasgow & Clyde
Locations (1):
- Children's Clinical Research Facility (CRF), Queen Elizabeth University Hospital, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hamilton R, Mulvihill A, Butler L, Chow A, Irving E, McCulloch DL, McNeil A, Michael K, Spowart KM, Waterson-Wilson J, Mactier H. Impaired vision in children prenatally exposed to methadone: an observational cohort study. Eye (Lond). 2024 Jan;38(1):118-126. doi: 10.1038/s41433-023-02644-3. Epub 2023 Jul 4. PMID 37402864